CLINICAL TRIAL: NCT05394363
Title: Generation Victoria Cohort 2020s. A Statewide Longitudinal Cohort of Victorian Children and Their Parents
Brief Title: Generation Victoria Cohort 2020s: A Statewide Longitudinal Cohort Study of Victorian Children and Their Parents
Acronym: GenV
Status: Recruiting | Type: Observational
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: The Paul Ramsay Foundation (Unknown); Royal Children's Hospital (Other); Victoria State Government (Unknown); Royal Children's Hospital Foundation (Unknown); University of Melbourne (Other); National Health and Medical Research Council, Australia (Other); Medical Research Future Fund (Other); Angliss Health Service (Unknown); Bairnsdale Regional Health Service (Unknown); Grampians Health - Ballarat Base Hospital (Unknown); Bass Coast Regional Health (Unknown); The Bays Private Hospital (Unknown); Benalla & District Memorial Hospital (Unknown); Bendigo Hospital (Unknown); Box Hill Hospital (Unknown); Cabrini Private Hospital (Unknown); Casey Hospital (Unknown); Castlemaine Hospital (Unknown); Central Gippsland Health Service (Unknown); Colac Area Health (Unknown); Dandenong Hospital (Unknown); Bacchus Marsh - Western Health (formerly Djerriwarrh Health Service) (Unknown); East Grampians Health Service (Unknown); Echuca Regional Health (Unknown); Epworth Freemason's Private Hospital (Unknown); Frances Perry Private Hospital (Unknown); Peninsula Health (Other Government); Epworth Geelong (Unknown); Geelong University Hospital (Unknown); Goulburn Valley Health (Unknown); Hamilton Base Hospital (Unknown); Jessie McPherson Private Hospital (Unknown); Joan Kirner Women's and Children's Hospital (Unknown); The Kilmore & District Hospital (Unknown); Latrobe Regional Hospital (Unknown); Leongatha Memorial Hospital (Unknown); Mansfield District Hospital (Unknown); Maryborough District Health Service (Unknown); Mercy Hospital for Women (Unknown); Mercy Werribee Public Hospital (Unknown); Mildura Base Hospital (Unknown); Mitcham Private Hospital (Unknown); Monash Medical Centre (Other); Northeast Health Wangaratta (Unknown); The Northern Hospital (Unknown); Northpark Private Hospital (Unknown); Peninsula Private Hospital (Unknown); Royal Women's Hospital (Unknown); Sandringham & District Memorial Hospital (Unknown); South Gippsland Hospital (Unknown); South West Healthcare Camperdown (Unknown); South West Healthcare Warnambool (Unknown); St John of God Hospital Ballarat (Unknown); St John of God Hospital Bendigo (Unknown); St John of God Hospital Berwick (Unknown); St John of God Hospital Geelong (Unknown); St Vincents Private Hospital (Unknown); Swan Hill District Hospital (Unknown); Waverley Private Hospital (Unknown); West Gippsland Healthcare Group (Unknown); Grampians Health - Horsham (formerly Wimmera Health Care Group) (Unknown); Albury Wodonga Health (Unknown); Yarrawonga District Health Service (Unknown); Portland District Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: U1111-1269-3107
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Mental Health; Child Wellbeing; Infant Health; Child Health; Reproductive Health; Healthy Aging; Health Equity; Quality of Life; Social Determinants of Health; Environmental Exposure; Genetics; Cognition; Learning; Child Development; Congenital Abnormalities; Disability; Injuries; Communicable Diseases; Noncommunicable Diseases; Physical Fitness; Diet; Obesity; Allergy and Immunology; Inflammation; Intergenerational Relations
Keywords: Generation Victoria; GenV; Cohort Studies; Data Collection; Data Linkage; Child Health; Midlife Health; Children; Infants; Family; Parents; Mothers; Fathers; Life course perspective; Population Health; Longitudinal Studies; Genetics, population; Demography; Epidemiology; Health Disparity; Minority Health; Vulnerable Populations; Health Equity; Clinical Trial; Randomized Controlled Trial; Pragmatic Clinical Trial; Health Services Research; Economic Models; Value of Life; Geographic Information Systems; Social Determinants of Health; Climate Change; Built Environment
MeSH Terms: conditions — Psychological Well-Being; Congenital Abnormalities; Wounds and Injuries; Communicable Diseases; Noncommunicable Diseases; Obesity; Hypersensitivity; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Universal residual biosamples from those already collected and stored by pathology providers:
  * Maternal Serum Screen (MSS) or Non-invasive Prenatal Test (NIPT)
  * Newborn Screening (NBS, Guthrie) cards
  * Prenatal biosamples from routine 1st, 2nd and 3rd trimester clinical pathology testing (eg. serum, whole blood and plasma throughout pregnancy, third trimester group B strep (GBS) vaginal/anal swab).
  New biosamples collected directly by GenV:
  * Saliva (child and parents)
  * Child stool
  * Breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Generation Victoria (GenV) is a longitudinal, population-based study of Victorian children and their parents that will bring together data on a wide range of conditions ,exposures and outcomes. GenV blends study-collected, study-enhanced and linked data. It will be multi-purpose, supporting observational, interventional, health services and policy research within the same cohort. It is designed to address physical, mental and social issues experienced during childhood, as well as the antecedents of a wide range of diseases of ageing. It seeks to generate translatable evidence (prediction, prevention, treatments, services) to improve future wellbeing and reduce the future disease burden of children and adults.

The GenV Cohort 2020s is open to all children born over a two-year period, and their parents, residing in the state of Victoria Australia. The GenV Cohort 2020s is preceded by an Advance Cohort of children born between 5 Dec 2020 and 3 October 2021, and their parents. This comprises all families recruited at GenV's Vanguard hospital (Joan Kirner Women's and Children's) and at birthing hospitals throughout Victoria as GenV scaled up to commence recruiting for the GenV Cohort 2020s. The Advance Cohort have ongoing and full participation in GenV for their lifetime unless they withdraw but may have less complete data and biosamples.

DETAILED DESCRIPTION:
GenV aims to create large, parallel whole-of-state birth and parent cohorts for discovery and interventional research. The four cornerstones of GenV's first decade are:

* Consented Cohort - Targeting all Victorian children born in a 2-year period and their parents, with the first major recruitment period targeting newborns and infants
* Biosamples - Curation of residual universal biosamples and collection of new biosamples
* Accessing existing data - Continuously-updated linkage to or ingestion of extensive administrative, service, geospatial and clinical datasets, including prospectively-collected datasets from before the child's birth
* Early School Wave - GenV-led phenomic assessment during the child's early school years.

Additional foundations activities are:

* GenV-collected survey data
* Integrated studies - Collaborative observational or interventional research studies embedded within or alongside GenV, with ethically-supported agreements that include arrangements for data sharing.
* IT and data platforms - to support all GenV activities including user research data access.

GenV focuses on 10 big issues: COVID, healthy pregnancy, healthy newborns, equity, climate & environment, mental health, healthy development, allergy & immunity, infection, and obesity & diabetes, with a cross cutting commitment of population genomics. These focus areas drive current planning for data collection but are not intended to be exhaustive and may change over the life of the project.

GenV partnered with all birthing hospitals across Victoria (i.e. 58 hospital sites). In-hospital face-to-face recruitment took place during the newborn period (December 2020 - November 2023). Recruitment visits were completed by trained study staff with clinical and/or research backgrounds, including initial GenV-collected data and biosamples. GenV remains open to eligible families through phone and/or self-guided recruitment.

Participant-provided data are collected digitally (e.g. via website or smart phone app) about four times per year from age 3 months to 1 year, then 6-12 monthly until 5 years, taking 3-20 minutes per session. A face-to-face visit is planned for when the index child is around 6-years of age, completed by trained study staff with clinical and/or research backgrounds. The project duration is expected to be at least 10 years and potentially lifelong for its participants, dependent on study funding and willingness to continue.

GenV estimated that the sampling frame for the main Cohort 2020s would comprise 150,000 children,150,000 birthing parents, and 130,000 (i.e. for 90 percent of children) second parents. GenV's recruitment rate is around 30% of all Victorian families with an eligible child. With a current sample size of 50,000 children, calculations show that this can detect odds ratios of around 1.3 for an outcome with 1.5% prevalence and an exposure with 20% prevalence.

ELIGIBILITY:
Inclusion Criteria (Children):

* Birth date between 4th October 2021 and 3rd October 2023
* Live at the time of recruitment
* Residing in Victoria at the time of recruitment
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the child's behalf, who provides a signed and dated informed consent form (e.g. a parent/guardian)

Inclusion Criteria (Adults):

* Be a parent or guardian of a child who meets the eligibility criteria above
* Provide a signed and dated informed consent form or have a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf.

Exclusion criteria:

* Children who are deceased at the time of recruitment (i.e. still born or died after birth) and their parents/guardians
* Families unable to provide informed consent in any of the languages available

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All children living in the state of Victoria, Australia, born between 4th October 2021 and 3rd October 2023, and their parents/guardians.
Sampling Method: Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2033-10 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Number of parents and children enrolled in the GenV Cohort 2020s | Point of consent until study completion (up to 10 years)
  Assessed by analysis of records in the study-specific Participant Relationship Management System (PRMS)
Number of participants with complete data collection at each wave | Point of consent until study completion (up to 10 years)
  Assessed by analysis of records in the study-specific Participant Relationship Management System (PRMS), e-Consent platform and GenV data repository
Number of participants with successful data linkage at each wave | Point of consent until study completion (up to 10 years)
  Assessed by analysis of records in the study-specific Participant Relationship Management System (PRMS), e-Consent platform and GenV data repository
Number of participants with the targeted biosamples received at each wave | Point of consent until study completion (up to 10 years)
  Assessed by analysis of records in the study-specific Participant Relationship Management System (PRMS), e-Consent platform and GenV Laboratory Information Management System (LIMS)

SECONDARY OUTCOMES:
Number of applications to access and analyse GenV end-user datasets | Point of consent until study completion (up to 10 years)
  Assessed by analysis of the GenV data access registry
Number of collaborative observational research studies supported | Point of consent until study completion (up to 10 years)
  Assessed by analysis of GenV Integrated Studies Register
Number of collaborative interventional research studies supported | Point of consent until study completion (up to 10 years)
  Assessed by analysis of GenV Integrated Studies Register
Number of participants involved in concurrent observational research studies embedded within or alongside GenV | Point of consent until study completion (up to 10 years)
  Assessed by analysis of shared study participant relationship management system data
Number of participants involved in concurrent interventional research studies embedded within or alongside GenV | Point of consent until study completion (up to 10 years)
  Assessed by analysis of shared study participant relationship management system data

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Wake, MBChB, FRACP, FAHMS, MD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Murdoch Children's Research Institute, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
GenV is designed as an Open Science resource. Privacy-protected child and parent research data will be made available spanning:
  * Individual physical and mental health, education, social and bioassay data
  * Neighbourhood data (eg pollution, childcare)
  Data will in general be made available after completion and data preparation for entire waves of data collection. An access policy is currently under development.
  GenV's biosamples are small in volume and depletable. Therefore, bioassay requests are most likely to proceed if they:
  * Are for all participants in GenV (or for the whole subgroup with that biosample)
  * Would be valued by many researchers
  * Generate broad, not hypothesis-specific, biodata (eg -omics panels)
  * Are supported by funding and quality processes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The first wave of data is expected to become publicly available in 2026. Subsequent releases will follow completed waves of data collection and are expected to be available indefinitely. Limited data are accessible to some collaborators prior to this, for example to support specific operations of integrated studies.
Access Criteria: Data will be made available to approved end-users for analyses that achieve the aims in the approved proposal. Approval is based on:
  * The research aims to improve health, development, or wellbeing
  * The proposed use of the data is covered by ethical approval
  * GenV assesses the safety and expertise of the applicant and the institution/organisation
  * Samples/data are used with participant privacy protection in place
  * Users agree to GenV's conditions of use.
URL: https://www.genv.org.au/for-researchers/enquire-about-collaborating-with-genv/

REFERENCES:
- [Derived] Hughes EK, Siero W, Gulenc A, Clifford SA, Frugier T, Hall SM, Mohal J, North K, Zaritski N, Goldfeld S, Saffery R, Wake M. Generation Victoria (GenV): protocol for a longitudinal birth cohort of Victorian children and their parents. BMC Public Health. 2025 Jan 3;25(1):20. doi: 10.1186/s12889-024-21108-1. PMID 39754130
- See also: Generation Victoria (GenV) Website — https://genv.org.au/
- Available data/document: GenV Protocol paper (open access) — https://doi.org/10.1186/s12889-024-21108-1 — Hughes, E.K., Siero, W., Gülenç, A. et al. Generation Victoria (GenV): protocol for a longitudinal birth cohort of Victorian children and their parents. BMC Public Health 25, 20 (2025).
- Available data/document: Informed Consent Form — https://doi.org/10.25374/MCRI.16902154 — Wake M, Goldfeld S, Saffery R; Siero W, Hughes E. Generation Victoria (GenV) Cohort 2020s Participant Information Statement and Consent Form In: Generation Victoria Figshare Project. Figshare 2021.
- Available data/document: Generation Victoria (GenV) Cohort 2020s Statement of Intent — https://doi.org/10.25374/MCRI.9962084 — Wake M, Goldfeld S, Saffery R, Siero W, Lamb K, Stringer M, et al. Generation Victoria (GenV) Cohort 2020s Statement of Intent In: Generation Victoria Figshare Project. Figshare 2019.
- Available data/document: Generation Victoria (GenV) Cohort 2020s Synopsis — https://doi.org/10.25374/MCRI.9122522 — Wake M, Goldfeld S, Saffery R, Siero W, Hourani D, Gulenc A, et al. Generation Victoria (GenV) Cohort 2020s Synopsis In: Generation Victoria Figshare Project. Figshare 2019.
- Available data/document: Guidance and expressions of interest for enquires and proposals to collaborate with GenV — https://genv.org.au/for-researchers/enquire-about-collaborating-with-genv/
- Available data/document: Current GenV collaborations — https://www.genv.org.au/for-researchers/current-genv-collaborations/
- Available data/document: Working Papers relevant to GenV design, data sharing and researchers working with GenV — https://genv.org.au/for-researchers/working-papers/
- Available data/document: Published Papers relevant to GenV design, data sharing and researchers working with GenV — https://genv.org.au/for-researchers/published-papers/